CLINICAL TRIAL: NCT02612012
Title: Phase II Study of Axillary Level I-II Areas Radiotherapy for Early Stage Breast Cancer With Limited Positive Sentinel Lymph Nodes
Brief Title: Axillary Radiotherapy for Early Stage Breast Cancer With Limited Positive Sentinel Lymph Nodes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Professor of department of radiation oncology, Fudan University
Other Study IDs: FDRT-BC002
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; positive sentinel lymph nodes; axillary radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Axillary radiotherapy
  Interventions: Radiation: axillary radiotherapy

INTERVENTIONS:
Radiation: axillary radiotherapy — Whole breast irradiation and axillary level I-II areas radiotherapy. The prescription dose is 50Gy in 25 fractions in 5 weeks. Tumor bed boost is necessary with 10Gy in 5 fractions in one week.

SUMMARY:
This study is designed to evaluate the feasibility and safety of axillary radiotherapy for early stage breast cancer with limited positive sentinel lymph nodes.

DETAILED DESCRIPTION:
Randomized clinical trials have demonstrated that complete axillary lymph node dissection is not necessary in patients with 1-2 positive sentinel lymph nodes who undergo breast conserving surgery, whole breast irradiation, and systemic therapy. However, whether or not the regional lymph node should be irradiated and if radiation given, whether or not all levels of axillary lymph node and internal mammary and supraclavicular lymph node should be irradiated is unknown. The purpose of this study is to evaluate the feasibility and safety of axillary level I-II areas radiotherapy for early stage breast cancer with 1-2 positive sentinel lymph nodes and no further axillary lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18~70 years old
* Pathologically confirmed invasive breast cancer
* A clinical T1-2N0M0 tumor
* Treated with breast conserving surgery and sentinel lymph node biopsy
* 1~2 positive sentinel lymph nodes, including micro-metastases or macro-metastases.
* ECOG score 1~2
* Written informed consent

Exclusion Criteria:

* Patients underwent complete axillary lymph node dissection
* Patients underwent mastectomy
* Patients underwent neoadjuvant therapy
* Clinically node positive pre-operative
* Sentinel lymph nodes only containing isolated tumour cells (<0.2 mm)
* Prior history of invasive breast cancer or previous or concurrent other malignancies within the past 5 years
* Previous radiation therapy of breast or thorax
* Medical contraindication for radiotherapy
* Prior axillary surgery or radiotherapy
* Unable or unwilling to receive breast conserving surgery or sentinel lymph node biopsy
* Pregnant or nursing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage breast cancer patients with 1~2 positive sentinel lymph nodes
Sampling Method: Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Axillary recurrence | 5 years

SECONDARY OUTCOMES:
Local-regional recurrence | 5 years
Disease free survival | 5 years
Overall survival | 5 years
Complications | baseline，1，2，3，4，5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD.PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China